CLINICAL TRIAL: NCT02451618
Title: A Pilot Study of Seizure Detection in Neonates Using Multimodal Temporary Epidermal Electronics
Brief Title: Novel Epidermal Recording and Detection of Seizures
Acronym: NERDS
Status: Terminated | Type: Observational
Why Stopped: Trial was discontinued due to inadequate signal from study eeg leads.
Sponsor: Sharp HealthCare (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, M J Harbert, Director of Neonatal Neurology, Sharp HealthCare
Other Study IDs: Epidermal Electronics
Record Dates: First submitted 2015-03-31; First posted 2015-05-22 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Seizures; Encephalopathy; Asphyxiated Newborn
Keywords: Perinatal Depression
MeSH Terms: conditions — Seizures; Brain Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Epidermal Electronic System: EES, wireless tattoo electrode
- Hydrogel electrode: EKG electrode, looking at hairline placement of electrodes.

SUMMARY:
For any newborn that exhibits possible seizure activity or has altered mental status of unknown etiology, continuous bedside EEG recording is the standard of care to detect subclinical seizure activity. The experimental aspect of this study will be the application of test electrodes (EES or EKG) to evaluate if the electrodes can be used to produce a continuous bedside recording of brain activity in the same manner as an EEG recording, while ideally producing less irritation of newborn skin than conventional EEG electrodes.

DETAILED DESCRIPTION:
Infants admitted to our NICU that require a standard EEG for clinical diagnosis will be approached for consent to test one of two new methods of EEG recording. Patients will be randomized to the new epidermal electronic system (EES) or the a hydrogel EKG electrode. All patients will continue to receive the standard of care EEG monitoring.

EES is slim new temporary tattoo technology that can easily be applied to the skin without requiring a technician or scrubbing and preparation as with standard EEG lead. The hydrogel EKG are FDA approved leads normally used to detect cardiac rhythm.

Specific Aims:

1. To compare the rate of detection of neonatal seizures between a new method of recording electrical brain rhythms (EES or EKG) and the current standard of care (EEG, or electroencephalography.)
2. To compare characterization of electrical brain activity between EES or EKG and EEG in the neonate.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized neonates who already require continuous EEG recording for clinical care
* Parents signed informed consent
* CGA 44 weeks or less

Exclusion Criteria:

* Patient is moribund

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any newborn admitted to the NICU that requires an EEG for clinical care. Must be less than or equal to 44 weeks corrected gestational age.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
Seizure detection | 24 hours
  Seizures detected by study electrodes will be compared to seizures detected on conventional EEG recording.

SECONDARY OUTCOMES:
EEG characterization | 24 hours
  Compare quality of brain activity with study leads vs standard leads
Skin integrity from standard EEG vs study electrodes | 24 hours
  Photographs will be taken to compare skin integrity after each electrode use.
Hair removal from standard EEG vs study electrodes | 24 hours
  If hair removal is necessary for study electrode placement.

OTHER OUTCOMES:
Apgar scores | Birth to 10 minutes of life
  Apgars at 1, 5, 10, 15, and 20 minutes of life if applicable
Subject received hypothermia treatment within 6 hours of life | Within 6 hours of life for 72 hours duration
Cause of seizure if known | Participants will be followed for the duration of hospital stay, an average of 10 days.
  Date and time of seizures and etiology
Anticonvulsant medication(s) subject received | Participants will be followed for the duration of hospital stay, an average of 10 days.
  Phenobarbital, Levetiracetam, Phosphenytoin, Versed, Blinded Study Drug, Other
Gestational age | At birth

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Harbert, MD, Principal Investigator — Sharp Mary Birch Hospital for Women & Newborns
Locations (1):
- Sharp Mary Birch Hospital for Women and Newborns, San Diego, California, United States

REFERENCES:
- [Background] Tharp BR. Neonatal seizures and syndromes. Epilepsia. 2002;43 Suppl 3:2-10. doi: 10.1046/j.1528-1157.43.s.3.11.x. PMID 12060001
- [Background] Lawrence R, Inder T. Neonatal status epilepticus. Semin Pediatr Neurol. 2010 Sep;17(3):163-8. doi: 10.1016/j.spen.2010.06.010. PMID 20727485
- [Background] Isaeva E, Isaev D, Savrasova A, Khazipov R, Holmes GL. Recurrent neonatal seizures result in long-term increases in neuronal network excitability in the rat neocortex. Eur J Neurosci. 2010 Apr;31(8):1446-55. doi: 10.1111/j.1460-9568.2010.07179.x. Epub 2010 Apr 6. PMID 20384780
- [Background] van Rooij LG, Toet MC, van Huffelen AC, Groenendaal F, Laan W, Zecic A, de Haan TR, van Straaten IL, Vrancken S, van Wezel G, van der Sluijs J, Ter Horst H, Gavilanes D, Laroche S, Naulaers G, de Vries LS. Effect of treatment of subclinical neonatal seizures detected with aEEG: randomized, controlled trial. Pediatrics. 2010 Feb;125(2):e358-66. doi: 10.1542/peds.2009-0136. Epub 2010 Jan 25. PMID 20100767
- [Background] Nagarajan L, Ghosh S, Palumbo L. Ictal electroencephalograms in neonatal seizures: characteristics and associations. Pediatr Neurol. 2011 Jul;45(1):11-6. doi: 10.1016/j.pediatrneurol.2011.01.009. PMID 21723453
- [Background] Ferree TC, Luu P, Russell GS, Tucker DM. Scalp electrode impedance, infection risk, and EEG data quality. Clin Neurophysiol. 2001 Mar;112(3):536-44. doi: 10.1016/s1388-2457(00)00533-2. PMID 11222977
- [Background] Young GB, Campbell VC. EEG monitoring in the intensive care unit: pitfalls and caveats. J Clin Neurophysiol. 1999 Jan;16(1):40-5. doi: 10.1097/00004691-199901000-00003. PMID 10082090
- [Background] Kim DH, Lu N, Ma R, Kim YS, Kim RH, Wang S, Wu J, Won SM, Tao H, Islam A, Yu KJ, Kim TI, Chowdhury R, Ying M, Xu L, Li M, Chung HJ, Keum H, McCormick M, Liu P, Zhang YW, Omenetto FG, Huang Y, Coleman T, Rogers JA. Epidermal electronics. Science. 2011 Aug 12;333(6044):838-43. doi: 10.1126/science.1206157. PMID 21836009
- [Background] Volpe JJ. Neonatal Seizures in Neurology of the Newborn, 4th ed. Philadelphia: WB Sanders, 2001: 178-214.